CLINICAL TRIAL: NCT03071887
Title: Developing a Resilience Intervention for Older, HIV-Infected Women
Brief Title: Resilience Intervention for Older, HIV-Infected Women
Acronym: BRIgHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Christina Psaros, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017P000404; R34AT009170 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-03-07 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Resilience, Psychological

STUDY DESIGN:
Intervention Model Description: This is an open pilot of the adapted Relaxation Response Resiliency Program (3RP).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Treatment arm - Relaxation Response Resiliency Program (3RP) (this is an open pilot; the treatment arm is the only arm)
  Interventions: Behavioral: Relaxation Response Resiliency Program (3RP)

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program (3RP) — The 3RP blends stress management principles, cognitive behavioral therapy, and positive psychology. The 3RP focuses on 3 major areas: (1) eliciting the relaxation response; (2) increasing stress awareness; and (3) promoting adaptive strategies. The 3RP intervention currently consists of eight, 90-minute weekly group sessions. The investigators plan to adapt the intervention to address common concerns for older, HIV-infected women, including: stress of managing a chronic long-term, life threatening illness; additional medical comorbidities; pain and fatigue; stigma and social isolation; depression and anxiety; and sexuality concerns.

SUMMARY:
The goal of this study is to refine and pilot the Relaxation Response Resiliency (3RP) intervention for women age 50 and over who are living with HIV, a group especially burdened by stressors related both to aging and living with chronic disease. The investigators will adapt the 3RP resiliency intervention to the needs of this population and conduct preliminary testing of the group intervention via an open pilot study.

DETAILED DESCRIPTION:
Overview.

Participants will be women living with HIV (N=up to 40) age 50 or over. Women will be recruited from the Boston area. Based on the investigators' qualitative work, the investigators will deliver an adapted version of the 3RP resiliency intervention to groups of 5-8 HIV-infected women age 50 and over. The 3RP intervention will consist of 8-10 weekly sessions of 90 minutes each focused on skills training to build and enhance resilience. The investigators will conduct baseline and post-treatment quantitative assessments, in addition to individual exit interviews to solicit feedback on the intervention. These data will be used to inform the design of a future randomized pilot study.

Study procedures.

Participants (N = up to 40) will be HIV-infected women age 50 or over . Participants will be recruited via study flyers (posted in the infectious disease clinics at local hospitals and in the waiting areas of Boston area community organizations) and provider referral. Once an individual expresses interest in the study, a research assistant will screen that individual to assess study eligibility criteria. Individuals who meet inclusion criteria will be invited to sign informed consent and complete an in-person baseline assessment. Participants will then complete the intervention (described below), a post-treatment assessment, and an individual in-depth exit interview to provide feedback on their experience in the study.

3RP Intervention:

Once enrolled in the study, participants will complete weekly group sessions of the 3RP intervention. Sessions will focus on developing an understanding of stress sources and physiology, and on developing a regular practice of eliciting the relaxation response (RR) and learning cognitive behavioral and positive psychology skills to enhance resiliency to long-term stress. Participants will be encouraged to practice skills (RR practice, thoughts records to learn adaptive thinking) between group sessions.

ELIGIBILITY:
Inclusion Criteria:

* biologically born women who endorse a female identity
* HIV-infected
* age 50 or older
* English speaking

Exclusion Criteria:

* presence of an active (i.e. untreated) and interfering psychiatric disorder (e.g., bipolar disorder, schizophrenia, substance abuse)
* have participated in a structured cognitive behavioral therapy and/or a mind-body intervention in the past year

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators will recruit biologically born women who endorse a female gender identity.
Enrollment: 13 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Psaros, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanton AM, Goodman GR, Blyler A, Kirakosian N, Labbe AK, Robbins GK, Park ER, Psaros C. Mental Health, Social Connectedness, and Fear During the COVID-19 Pandemic: A Qualitative Perspective from Older Women with HIV. AIDS Behav. 2023 Jul;27(7):2176-2189. doi: 10.1007/s10461-022-03950-9. Epub 2022 Dec 20. PMID 36538139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The three open pilot groups and qualitative exit interviews were conducted between December 2017 and July 2018 through community outreach, flyers, and referrals from healthcare providers at the Infectious Disease units of two Boston-area hospitals.
Groups:
- Treatment: Relaxation Response Resiliency Program (3RP): The 3RP blends stress management principles, cognitive behavioral therapy, and positive psychology. The 3RP focuses on 3 major areas: (1) eliciting the relaxation response; (2) increasing stress awareness; and (3) promoting adaptive strategies. The 3RP intervention currently consists of eight, 90-minute weekly group sessions. The investigators adapted the intervention to address common concerns for older, HIV-infected women, including: stress of managing a chronic long-term, life threatening illness; additional medical comorbidities; pain and fatigue; stigma and social isolation; depression and anxiety; and sexuality concerns.
Period: Overall Study
Arm/Group | Treatment: Relaxation Response Resiliency Program (3RP)
Started | 13
Completed | 7
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: Relaxation Response Resiliency Program (3RP)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 8
  White | 4
  Other | 1
Education [Count of Participants; unit: Participants]
  Less than high school degree | 5
  High school graduate/GED | 1
  College/graduate school partial/degree | 7
Current Employment Status [Count of Participants; unit: Participants]
  Full-Time | 1
  Part-Time | 2
  Disabled/retired | 9
  Other | 1
Relationship Status [Count of Participants; unit: Participants]
  Single | 5
  Married/Partnered | 3
  Separated/Divorced | 5
Monthly Income [Count of Participants; unit: Participants]
  $10,000 or less | 9
  More than $10,000 | 4
Years since diagnosis [Count of Participants; unit: Participants]
  More than 5 years ago | 12
  Less than 5 years ago | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Treatment Sessions
Description: The investigators will assess feasibility by collecting data on the number of completed treatment sessions.
Time Frame: Approximately 10 weeks after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Relaxation Response Resiliency Program (3RP)
Number analyzed (Participants) | 13
Participants
  Attended at least half of group sessions | 4
  Attended fewer than half of group sessions | 9

2. Primary Outcome: Participant Satisfaction With Study Procedures
Description: Acceptability will be assessed using scores on the Client Satisfaction Questionnaire (CSQ-8). Response options as follows, "Very satisfied", "Mostly satisfied", "Indifferent or mildly dissatisfied", and "Quite dissatisfied".
Time Frame: Approximately 10 weeks after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Relaxation Response Resiliency Program (3RP)
Number analyzed (Participants) | 7
Participants
  Very satisfied | 6
  Mostly satisfied | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 8 months study enrollment and participation (December 2017 through August 2018).
Arm/Group | Treatment: Relaxation Response Resiliency Program (3RP)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03071887/Prot_SAP_000.pdf